CLINICAL TRIAL: NCT02149290
Title: LifeVest Trends Validation Protocol
Acronym: TRENDS
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90D0120
Record Dates: First submitted 2014-05-01; First posted 2014-05-29 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; Six minute walk test
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Trends-equipped LifeVest 4000: Subjects using the LifeVest 4000 modified to collect Trends data
  Interventions: Device: Trends-equipped LifeVest 4000

INTERVENTIONS:
Device: Trends-equipped LifeVest 4000 — LifeVest 4000 monitors patients for VT/VF, notifies the patient if VT/VF occurs, and instructs them to press response buttons. In unresponsive patients, LifeVest delivers defibrillation therapy. Trends modifications for heart failure monitoring include: body position data collection; heart rate measurements, activity data collection; ability to perform a health survey; ability to guide patients through a walk test

SUMMARY:
This study will evaluate the accuracy of data on body position, daily activity, heart rate, 6-minute walk test, and a health survey collected by the wearable cardioverter defibrillator (WCD).

DETAILED DESCRIPTION:
This is a multi-center validation study of heart failure patients wearing the LifeVest WCD modified to collect data on body position, activity, heart rate, 6-minute walk test, and a health survey in order to evaluate data accuracy and patient interactions with the device.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic heart failure (i.e., New York Heart Association (NYHA) class II or higher)
* Evidence of a prior Myocardial Infarction (MI) or dilated cardiomyopathy
* Ejection fraction of 35% or less at the start of WCD use
* Anticipated to need a WCD for three months or more
* At least 18 years of age (over the legal age of providing consent)

Exclusion Criteria:

* Use of an implantable cardioverter defibrillator (ICD), recent removal of an ICD, or planned use of an ICD within the next three months
* Need for an assistive device for ambulation (wheelchair, walker, or cane)
* Use of a unipolar pacemaker
* Physical or mental conditions that prevent interaction with or wearing of the device
* Advanced directive prohibiting resuscitation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure who are being cared for in an outpatient environment
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2014-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Szymkiewicz, MD, Study Director — Zoll Medical Corporation
Locations (21):
- United States (13):
  - Orange County Heart Institute, Orange, California
  - Cardiac Arrhythmia Service, Boca Raton, Florida
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Lexington Cardiology Consultants, Lexington, Kentucky
  - Cardiology Institute of Michigan, Flint, Michigan
  - SUNY Downstate, Brooklyn, New York
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Erlanger Clinical Research, Chattanooga, Tennessee
  - Methodist Healthcare Foundation, Memphis, Tennessee
  - VA Beach General, Virginia Beach, Virginia
  - Swedish Medical Center, Seattle, Washington
  - CAMC, Charleston, West Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
- Klinische Abteilung für Kardiologie, Graz, Austria
- Germany (7):
  - Universitats-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Kerckhoff-Klinik, Bad Nauheim
  - Medizinische Klinik & Poliklinik II - Kardiologie, Bonn
  - Klinikum Coburg, Coburg
  - St. Vinzenz Hospital, Cologne
  - Department für Herzinsuffizienz und Devicetherap, Hamburg
  - Klinik für Innere Medizin III, Villingen-Schwenningen

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trends-equipped LifeVest 4000
Started | 198
Completed | 198
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Trends-equipped LifeVest 4000
Number analyzed (Participants) | 198
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 151
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 27
  United States | 81
  Germany | 90
Baseline Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: Ejection Fraction Percentage] | 23 (7)
New York Heart Association Classification [Count of Participants; unit: Participants] — Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  No NYHA class listed or unable to determine.
  Participants
    Class I | 0
    Class II | 102
    Class III | 83
    Class IV | 11
    Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Distance Traveled in Six Minute Walk Test
Description: Relationship of the step count and distance measure of the LifeVest walk test in heart failure patients as compared to distance measure of medically supervised 6-minute walk test. Accuracy of activities, and body position in patients with heart failure as compared to patient diaries of activity and sleeping position.
Time Frame: Three months
Population: All participants that had at least one recorded in-clinic 6MWT
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Clinician Guided 6MWT: Distance-First Clinician guided 6MWT
- WCD Guided 6MWT: Distance-First WCD guided 6MWT
Arm/Group | Clinician Guided 6MWT | WCD Guided 6MWT
Number analyzed (Participants) | 100 | 78
meters | 306 (100) | 296 (100)

2. Secondary Outcome: Compliance With Completing 6MWT Through a Wearable Defibrillator.
Description: Observe Compliance with completing weekly 6MWT
Time Frame: Up to 12-14 Weeks of WCD use
Population: All participants
Measure: Number; unit: % of participants completing >= 1 6MWT
Arm/Group | Trends-equipped LifeVest 4000
Number analyzed (Participants) | 198
% of participants completing >= 1 6MWT | 79

3. Secondary Outcome: Observe Compliance With Answering Questions Regarding Health Through a Wearable Defibrillator.
Description: Observe compliance with answering daily health survey.
Time Frame: Up to 12-14 Weeks of WCD use
Population: All participants.
Measure: Number; unit: % of participants completing >= 1 survey
Arm/Group | Trends-equipped LifeVest 4000
Number analyzed (Participants) | 198
% of participants completing >= 1 survey | 93

4. Other Pre Specified Outcome: Patient Interactions With the Wearable Defibrillator
Description: Compliance with WCD use during the study period, and patient-device interactions during a ventricular arrhythmia, if any should occur during the study period.
Time Frame: Three months
Population: All participants
Measure: Median (Inter-Quartile Range); unit: Days worn
Arm/Group | Trends-equipped LifeVest 4000
Number analyzed (Participants) | 198
Days worn | 78 [45.5 to 98.5]

ADVERSE EVENTS:
Time Frame: During the 12-14 weeks of WCD use
Description: All adverse events during the study period whether or not considered related to the participant's participation in the research.
Arm/Group | Trends-equipped LifeVest 4000
All-Cause Mortality (participants affected / at risk) | 0/198
Serious Adverse Events (participants affected / at risk) | 5/198
Other Adverse Events (participants affected / at risk) | 0/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trends-equipped LifeVest 4000 (N=198)
Tachycardia (Cardiac disorders) | 3 (4)
Dyspnea (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT02149290/Prot_SAP_000.pdf